CLINICAL TRIAL: NCT06948747
Title: An Open-label, Fixed-sequence, Three-part Study to Assess the Effect of AZD5004 on the Pharmacokinetics of Rosuvastatin, Atorvastatin, Simvastatin, Repaglinide and to Assess the Effect of Erythromycin on AZD5004 in Healthy Participants
Brief Title: A Study to Investigate the Effect of AZD5004 on Rosuvastatin, Atorvastatin, Simvastatin, Repaglinide and the Effect of Erythromycin on AZD5004 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: D7260C00017
Record Dates: First submitted 2025-04-28; First posted 2025-04-29 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: Obesity; Type 2 Diabetes Mellitus (T2DM); Pharmacokinetics
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Rosuvastatin Calcium; Erythromycin; Atorvastatin; Simvastatin; repaglinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): Participants will receive 10 mg rosuvastatin in Period 1. Participants will receive 10 mg rosuvastatin and AZD5004 in Period 2. Later, participants will receive different doses of AZD5004 followed by 10 mg single dose of rosuvastatin in Period 3, Period 4, Period 5, and Period 6. In Period 7, participants will receive AZD5004 alone and later, 500 mg erythromycin twice a day. Participants will receive 500 mg erythromycin co-administered with AZD5004 during Period 8.
  Interventions: Drug: AZD5004; Drug: Rosuvastatin; Drug: Erythromycin
- Part B (Experimental): Participants will receive 20 mg simvastatin during Period 1. In Period 2, participants will receive 40mg atorvastatin. In Period 3, participants will receive 40 mg atorvastatin and then, AZD5004 once daily . During Period 4, participants will receive 40 mg atorvastatin with single dose of AZD5004 and later, two different doses of AZD5004 alone will be administered once a day. In Period 5, participants will receive 20 mg simvastatin with single dose of AZD5004, later, AZD5004 alone will be administered once a day. During Period 6, participants will receive 40 mg atorvastatin with single dose of AZD5004 initially, and later AZD5004 will be administered once daily. In Period 7, participants will receive AZD5004 followed by 40 mg single dose of atorvastatin.
  Interventions: Drug: AZD5004; Drug: Atorvastatin; Drug: Simvastatin
- Part C (Experimental): Participants will receive 0.5 mg repaglinide initially during Period 1, later AZD5004 once daily will be administered . Participants will then receive 0.5 mg repaglinide with single dose of AZD5004 in Period 2, later two different doses of AZD5004 once daily will be administered. In Period 3, participants will receive 0.5 mg repaglinide with single dose of AZD5004 initially, and later AZD5004 once daily will be administered. In Period 4, participants will receive 0.5 mg repaglinide with single dose of AZD5004.
  Interventions: Drug: AZD5004; Drug: Repaglinide

INTERVENTIONS:
Drug: AZD5004 — Participants will receive oral tablets of AZD5004 as single dose on the following days, (i) Day 7, Day 14, Day 21, Day 28, Day 35, Day 42 and Day 55 in Part A. (ii) Day 9 to Day15, Day 16, Day 17 to Day 23, Day 24 to Day 30, Day 31 to Day 37, Day 38 to Day 41 and Day 42 in Part B.
  (iii) Day 3 to Day 9, Day 10 to Day 25, Day 26 to Day 33, and Day 34 in Part C.
Drug: Rosuvastatin — Participants will receive single oral tablets of rosuvastatin 10mg on Days 1, 7, 14, 21, 28, and 35.
  Arms: Part A
Drug: Erythromycin — Participants will receive oral doses of erythromycin 500 mg, twice a day from Day 49 to Day 54; and a single dose of 500 mg on Day 55.
  Arms: Part A
Drug: Atorvastatin — Participants will receive single oral doses of 40 mg atorvastatin on Days 4, 8, 16, 38, and 42.
  Arms: Part B
Drug: Simvastatin — Participants will receive single oral doses of 20 mg simvastatin on Days 1 and 31.
  Arms: Part B
Drug: Repaglinide — Participants will receive single oral doses of 0.5 mg repaglinide on Days 1, 10, 26, and 34.
  Arms: Part C

SUMMARY:
This study will assess the effect of AZD5004 on Rosuvastatin, Atorvastatin, Simvastatin, Repaglinide and the effect of Erythromycin on AZD5004 in healthy adult male and female participants.

DETAILED DESCRIPTION:
This is a Phase I, open-label, fixed-sequence, single center study which consists of 3 parts: Part A, Part B and Part C. Part A, Part B, and Part C are 3 independent and non-sequential parts in this study.

The purpose of Part A (Rosuvastatin and Erythromycin) of this study is to measure the following in healthy male and female participants,

1. The impact of AZD5004 on the pharmacokinetics (PK: the way the body absorbs, distributes, metabolizes, and eliminates a medicine) of rosuvastatin and
2. The impact of erythromycin on the PK of AZD5004

The purpose of Part B (Atorvastatin and Simvastatin) of this study is to measure the impact of AZD5004 on the PK of atorvastatin and simvastatin in healthy male and female participants.

The purpose of Part C (Repaglinide) of this study is to measure the impact of AZD5004 on the PK of repaglinide in healthy male and female participants.

Part A will consist of a screening period, 8 treatment periods, and a follow-up period.

Part B will consist of a screening period, 7 treatment periods, and a follow-up period.

Part C will consist of a screening period, 4 treatment periods, and a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged 18 to 55 years
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Female(s) of childbearing potential if heterosexually active, must agree to use an approved method of highly effective contraception.
* Male participants must use condoms for the duration of clinical trial.
* Additional contraception must be used for the sexual partners of male trial participants throughout the clinical trial.
* Have a body mass index (BMI) between ≥ 20.0 and ≤ 35 kg/m2 (at the time of screening) inclusive and weigh at least 50 kg.

Exclusion Criteria:

* History of any clinically important disease or disorder (liver transplant, liver disease, positive for serum HBsAg (Hepatitis B surface antigen) OR anti-HBcAb (Hepatitis B core antibody), positive for anti-HCV (Hepatitis C virus), history of cirrhosis and/or hepatic decompensation, cardiovascular disease, neuromuscular or neurogenic disease.
* History of Type 1 or Type 2 diabetes mellitus (DM).
* History of Hemoglobin A1c ≥ 6.5% (≥ 48 mmol/mol) at screening.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma.
* Any laboratory values with deviations or clinically important abnormalities in clinical chemistry, hematology, or urinalysis at the Screening Visit or on admission to the Clinical Unit.
* Significant hepatic disease as judged by the investigator.
* Any positive result on screening for serum HBsAg, HBcAb or HIV (Human immunodeficiency virus).
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12 lead ECG, at screening
* Abnormal vital signs.
* Uncontrolled thyroid disease or history/family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2).
* Current smokers or those who have smoked or used nicotine products.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the investigator. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for females.
* Positive screen for drugs of abuse, or alcohol or cotinine at screening or on each admission to the Clinical Unit.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Excessive intake of caffeine-containing drinks or food
* History of psychosis or bipolar disorder or major depressive disorder or suicide attempt or suicidal ideation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Part A, Part B and Part C: Area under concentration time curve from time 0 to infinity (AUCinf) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the effect of single dose of AZD5004 on the PK of a single dose of rosuvastatin and multiple doses of erythromycin on the PK of a single dose of AZD5004 in healthy participants.
  Part B: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of atorvastatin and atorvastatin metabolites (o-hydroxy atorvastatin and p-hydroxy atorvastatin) and simvastatin and simvastatin metabolites (simvastatin acid) in healthy participants.
  Part C: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of repaglinide in healthy participants.
Part A, Part B and Part C: Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the effect of single dose of AZD5004 on the PK of a single dose of rosuvastatin and multiple doses of erythromycin on the PK of a single dose of AZD5004 in healthy participants.
  Part B: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of atorvastatin and atorvastatin metabolites (o-hydroxy atorvastatin and p-hydroxy atorvastatin) and simvastatin and simvastatin metabolites (simvastatin acid) in healthy participants.
  Part C: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of repaglinide in healthy participants.
Part A, Part B and Part C: Maximum observed drug concentration (Cmax) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the effect of single dose of AZD5004 on the PK of a single dose of rosuvastatin and multiple doses of erythromycin on the PK of a single dose of AZD5004 in healthy participants.
  Part B: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of atorvastatin and atorvastatin metabolites (o-hydroxy atorvastatin and p-hydroxy atorvastatin) and simvastatin and simvastatin metabolites (simvastatin acid) in healthy participants.
  Part C: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of repaglinide in healthy participants.
Part A, Part B and Part C: Terminal elimination half life (t½λz) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the effect of single dose of AZD5004 on the PK of a single dose of rosuvastatin and multiple doses of erythromycin on the PK of a single dose of AZD5004 in healthy participants.
  Part B: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of atorvastatin and atorvastatin metabolites (o-hydroxy atorvastatin and p-hydroxy atorvastatin) and simvastatin and simvastatin metabolites (simvastatin acid) in healthy participants.
  Part C: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of repaglinide in healthy participants.
Part A, Part B and Part C: Terminal rate constant (λz) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the effect of single dose of AZD5004 on the PK of a single dose of rosuvastatin and multiple doses of erythromycin on the PK of a single dose of AZD5004 in healthy participants.
  Part B: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of atorvastatin and atorvastatin metabolites (o-hydroxy atorvastatin and p-hydroxy atorvastatin) and simvastatin and simvastatin metabolites (simvastatin acid) in healthy participants.
  Part C: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of repaglinide in healthy participants.
Part A, Part B and Part C: Time to reach maximum observed concentration (tmax) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the effect of single dose of AZD5004 on the PK of a single dose of rosuvastatin and multiple doses of erythromycin on the PK of a single dose of AZD5004 in healthy participants.
  Part B: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of atorvastatin and atorvastatin metabolites (o-hydroxy atorvastatin and p-hydroxy atorvastatin) and simvastatin and simvastatin metabolites (simvastatin acid) in healthy participants.
  Part C: To assess the effect of multiple doses of AZD5004 on the PK of a single dose of repaglinide in healthy participants.
Part A, Part B and Part C: Ratio Area under concentration time curve from time 0 to infinity (RAUCinf) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the Ratio of Rosuvastatin (Rosuvastatin + AZD5004) to Rosuvastatin (alone) and Ratio of AZD5004 (AZD5004 + erythromycin) to AZD5004 (alone) based on AUCinf.
  Part B: To assess the Ratio of Atorvastatin or Simvastatin (Atorvastatin/Simvastatin + AZD5004) to Atorvastatin or Simvastatin (alone) based on AUCinf.
  Part C: To assess the Ratio of Repaglinide (Repaglinide + AZD5004) to Repaglinide (alone) based on AUCinf.
Part A, Part B and Part C: Ratio of Area under concentration curve from time 0 to the last quantifiable concentration (RAUClast) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the Ratio of Rosuvastatin (Rosuvastatin + AZD5004) to Rosuvastatin (alone) and Ratio of AZD5004 (AZD5004 + erythromycin) to AZD5004 (alone) based on AUClast.
  Part B: To assess the Ratio of Atorvastatin or Simvastatin (Atorvastatin/Simvastatin + AZD5004) to Atorvastatin or Simvastatin (alone) based on AUClast.
  Part C: To assess the Ratio of Repaglinide (Repaglinide + AZD5004) to Repaglinide (alone) based on AUClast.
Part A, Part B and Part C: Ratio of Maximum observed drug concentration (RCmax) | Part A:Days 1-4, 7-10, 14-17, 21-24, 28-31, 35-38, 42-49 and 55-62 Part B:Days 1, 2, 4-7, 8-11, 15, 16-19, 23, 24, 30, 31, 32, 37, 38-41, 42-45 Part C:Days 1, 2, 9, 10, 11, 18, 19, 25, 26, 27, 33, 34-36
  Part A: To assess the Ratio of Rosuvastatin (Rosuvastatin + AZD5004) to Rosuvastatin (alone) and Ratio of AZD5004 (AZD5004 + erythromycin) to AZD5004 (alone) based on Cmax.
  Part B: To assess the Ratio of Atorvastatin or Simvastatin (Atorvastatin/Simvastatin + AZD5004) to Atorvastatin or Simvastatin (alone) based on Cmax.
  Part C: To assess the Ratio of Repaglinide (Repaglinide + AZD5004) to Repaglinide (alone) based on Cmax.

SECONDARY OUTCOMES:
Part A, Part B and Part C: Number of participants with adverse events (AEs) and adverse event of special interest (AESI) | Part A: From screening (Day -28 to -2 ) to followup visit (Day 65) Part B: From screening (Day -28 to -2) to followup visit (Day 48) Part C: From screening (Day -28 to -2) to followup visit (Day 38)
  To examine the safety and tolerability of AZD5004 alone and in combination with, the following drugs in healthy participants as listed below Part A: rosuvastatin or erythromycin Part B: atorvastatin and simvastatin Part C: repaglinide

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/